CLINICAL TRIAL: NCT00787683
Title: Home-Monitoring in ICD Patients
Brief Title: Home-Monitoring in Implantable Cardioverter Defibrillator (ICD) Patients
Acronym: Monitor-ICD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: F. Mueller-Riemenschneider (Other)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor-Investigator, F. Mueller-Riemenschneider, PD, Dr., Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V7.0
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Ventricular Arrythmias
Keywords: Patients with ventricular arrhythmias and the prevention of sudden cardiac death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home-monitoring (Experimental): Patients receive an additional home-monitoring (remote-monitoring) device (CardioMessengerII) following Biotronik Lumax ICD implantation. The device enables regular transmission and examination of ICD information via home-monitoring. Follow-up appointments in outpatient clinic are changed compared to standard care. While follow-up 1, 12, and 24 months after ICD implantation consist of outpatient clinic appointments, follow-up 3, 6, and 18 months after ICD implantation are conducted remotely.
  Interventions: Device: Home-monitoring provided by LUMAX ICD device and CardioMessenger II
- Standard care (No Intervention): Patients randomised to the standard care group receive no home-monitoring device (CardioMessengerII) following Lumax ICD implantation. Patients have scheduled follow-up appointments at the ICD outpatient clinics at 1, 3, 6, 12, 18, and 24 months after ICD implantation.

INTERVENTIONS:
Device: Home-monitoring provided by LUMAX ICD device and CardioMessenger II — All study participants receive an ICD of the Biotronik lumax family. Only participants of the intervention group receive the CardioMessengerII to allow for transmission of regular home monitoring messages. All study participants will be followed for 12 to 24 months (depending on the time of recruitment). The intervention and comparison to be investigated is home-monitoring vs. no home-monitoring. The intervention involves a combination of in-clinic consultations and regular use of home-monitoring services. As part of the modified follow-up schedule of intervention patients compared to standard care, follow-up in-clinic consultations 3, 6, and 18 months after ICD implantation will be replaced by home-monitoring follow-up.
  Other Names: Home-monitoring; Remote-monitoring; Tele-monitoring; ICD; Biotronik; Lumax; CardioMessenger
  Arms: Home-monitoring

SUMMARY:
The purpose of this study is to investigate the cost-effectiveness and effectiveness of remote-monitoring compared to standard care in patients with implantable cardioverter defibrillator.

DETAILED DESCRIPTION:
Implantable cardioverter defibrillator (ICD) are an important and effective treatment in patients at risk of sudden cardiac death. In order to allow for a more continuous follow-up and reduced complication rates of patients with ICD, new devices including remote-monitoring (home-monitoring) features of patients with ICD have been developed. BIOTRONIK Home Monitoring service enables the doctors to safely follow up their patients with implanted cardioverter-defibrillators in a remote fashion, with fewer in-clinic consultations. This may result in a more efficient follow-up and cost-savings for the health care payer.

The objective of the current study is to investigate the cost-effectiveness and effectiveness of home-monitoring compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* The patient is willing/able to undergo the study protocol appointments and procedures/questionnaires
* Indication for implantation of single chamber ICD or dual chamber ICD according to European guidelines

Exclusion Criteria:

* Age < 18 and > 80 years
* Expected non-compliance
* Known drug or alcohol abuse
* Life expectancy < 1 year
* NYHA classification IV
* Participation in another clinical study
* Participation in another telemonitoring concept
* Pregnant or breast-feeding woman
* Uncontrolled hypertension
* No mobile phone use possible in patient residence

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2008-10; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of disease specific costs from a societal perspective. | up to 24 months

SECONDARY OUTCOMES:
Number of shocks | up to 24 months
Hospital admissions | up to 24 months
Cardiac events | up to 24 months
Quality of life | up to 24 months
Disease specific Costs from third party payers perspective | up 24 months
Overall costs from societal and third party payers perspective | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Markus Zabel, Prof., MD, Principal Investigator — Medical Faculty, University of Göttingen, Germany
Locations (13):
- Germany (13):
  - Asklepios Hospital Barmbeck in Hamburg, Hamburg, Hamburg
  - Hospital Bremerhaven, Bremerhaven, Lower Saxony
  - MH-Hannover, Hanover, Lower Saxony
  - University Hospital Aachen, Aachen, North Rhine-Westphalia
  - Cardiological Practice, Bonn, North Rhine-Westphalia
  - St. Vincenz Hospital Paderborn, Paderborn, North Rhine-Westphalia
  - University Hospital Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Hospital Bad Berka, Bad Berka
  - Hospital Coburg, Coburg
  - University Hospital Göttingen, Göttingen
  - Heart Centre Bodensee Konstanz, Konstanz
  - University Hospital Münster, Münster
  - Academic Teaching Hospital Villingen of the University of Freiburg, Villingen-Schwenningen

REFERENCES:
- [Derived] Zabel M, Muller-Riemenschneider F, Geller JC, Brachmann J, Kuhlkamp V, Dissmann R, Reinhold T, Roll S, Luthje L, Bode F, Eckardt L, Willich SN; MONITOR-ICD investigators. Rationale and design of the MONITOR-ICD study: a randomized comparison of economic and clinical effects of automatic remote MONITORing versus control in patients with Implantable Cardioverter Defibrillators. Am Heart J. 2014 Oct;168(4):430-7. doi: 10.1016/j.ahj.2014.04.021. Epub 2014 Jun 13. PMID 25262251